CLINICAL TRIAL: NCT02125474
Title: Efficacy of Peptide Receptor Radionuclide Therapy for Metastatic Inoperable Neuroendocrine Tumors Using 177-Lu-DOTA 0, Tyr 3 Octreotate
Brief Title: Efficacy of 177-Lu-DOTA 0, Tyr 3 Octreotate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia, Columbia (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C41030610-041
Record Dates: First submitted 2014-04-22; First posted 2014-04-29 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2014-05

CONDITIONS: Neuroendocrine Tumors
Keywords: Neuroendocrine Tumors; Lutetium; Treatment Outcome
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Lutetium-177; copper dotatate CU-64

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- [177Lu] DOTA-TATE (Experimental): We have designed a one-arm phase II prospective sequential clinical trial to assess the therapeutic efficacy of 177-Lu-[DOTA 0, Tyr 3] octreotate (177-Lu- DOTATATE) applied intravenously in three separate doses to patients with inoperable progressive WDNET.
  Interventions: Radiation: [177Lu] DOTA-TATE

INTERVENTIONS:
Radiation: [177Lu] DOTA-TATE — We have designed a one-arm phase II prospective sequential clinical trial to assess the therapeutic efficacy of 177-Lu-[DOTA 0, Tyr 3] octreotate (177-Lu- DOTATATE) applied intravenously in three separate doses to patients with inoperable progressive WDNET.

SUMMARY:
Well-differentiated neuroendocrine tumors (WDNETs) are uncommon neoplasms with an increasing number of new cases reported in the annual statistics of the Instituto Nacional de Cancerología (INC). The majority are advanced-stage presentations with limited chances of a complete surgical resection of the primary tumor, a clinical scenario where medical treatment options are also limited. In view of the characteristically defined expression of peptide receptors in WDNETs, radioactive molecular probes to target specific cellular receptors have been designed using radioisotopes with short range of penetration in tissues. We have designed a one-arm phase II prospective sequential clinical trial to assess the therapeutic efficacy of 177-Lu-[DOTA 0, Tyr 3] octreotate (177-Lu- DOTATATE) applied intravenously in three separate doses to patients with inoperable progressive WDNET. Selected patients matching inclusion criteria will be enrolled at the INC's Section of Endocrinology. Tumor response, treatment safety (side effects) and survival will be appraised. Data from clinical, biochemical and imaging follow-up will be periodically registered during treatment and until two years after the last infusion of 177Lu- DOTATATE. This phase II trial is justified because despite the fact that many preclinical and clinical studies have showed the potential usefulness of this novel palliative approach to treat patients with advanced-stage WDNETs there is a paucity of vigorous results to establish its efficacy as first-line treatment.

DETAILED DESCRIPTION:
The Investigators have designed a one-arm phase II prospective sequential clinical trial to assess the therapeutic efficacy of 177-Lu-[DOTA 0, Tyr 3] octreotate (177-Lu- DOTATATE) applied intravenously in three separate doses to patients with inoperable progressive WDNET.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inoperable gastroenteropancreatic neuroendocrine tumors.
* Histopathologic diagnosis confirmed at the Instituto Nacional de Cancerología.
* Somatostatin receptor-positive tumors with at least one site of abnormal focal uptake > liver physiologic uptake (3+) observed in a 99mTc-HYNIC-TOC scintigraphy practiced less than 6 months before treatment with 177Lu- DOTATATE.
* Karnofsky functional score > 60.
* Life expectancy > 3 months.
* Multiple inoperable metastatic sites.
* Patient voluntarily willing to participate in the trial.
* Hemoglobin (Hb) > 8.8 g/dl
* Leucocytes (Leu) > 2 x 103/µl
* Platelets (Plaq) > 80 x 103/µl
* Total Bilirrubin (BT) ≤ 3 times the upper limit of normal range. Serum albumin > 3 g/dl and normal prothrombin time.
* At least one measurable CT tumor lesion.
* Non-lactating woman with negative pregnancy blood test.
* Creatinine clearance > 40 ml/min and serum creatinine < 1.5 mg/dl and/or isotopic glomerular filtration rate > 50 ml/min.
* Test results should predate treatment by at least: blood test results ≤ 4 weeks, liver blood tests < 1 month, renal function tests < 1 week, CT ≤ 4 months and 99mTc-HYNIC-TOC scintigraphy < 6 months.

Exclusion Criteria:

* Patients previously treated with radionuclide therapy.
* Patients treated with chemo- o radiotherapy within the past 6 months.
* Patients unable to comply with clinical follow-up in both Nuclear Medicine and Endocrinology units.
* Patients unwilling to participate in the trial or not providing written informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Response to treatment | 3 years
  Response to palliative treatment with 177Lu- DOTATATE in patients with metastatic progressive low-grade neuroendocrine tumors defined by control size tumor, response time to reduction minimal parcial and complete tumor.

SECONDARY OUTCOMES:
Efficacy defined by reduction in size tumoral | 3 years
  Measure the efficacy of 177Lu- DOTATATE to treat patients with metastatic progressive low-grade neuroendocrine tumors using clinical and imaging criteria such as tumor size.
Side effects defined by clinical follow up | 5 years
  Describe the side effects of the treatment with 177Lu- DOTATATE by clinical follow-up during and after therapy
survival rate | 2 years
  describe the 2-year survival rate of patients treated with 177Lu- DOTATATE
Quality of life | 3 years
  Assess the quality of life of patients with metastatic progressive low-grade neuroendocrine tumors treated with 177Lu- DOTATATE during treatment defined by pain reduction and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen A De los Reyes, Md, Principal Investigator — Instituto Nacional de Cancerologia de Mexico
Locations (1):
- Instituto Nacional de Cancerología, Bogota, Cundinamarca, Colombia